CLINICAL TRIAL: NCT06078982
Title: Efficacy and Safety of Disitamab Vedotin Combined With PD-1 in Posterior Line Therapy of Advanced HER2-low Expressing Gastric Cancer
Brief Title: Posterior-line Treatment With Disitamab Vedotin Plus PD-1 in Advanced HER2-low Expressing Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Jin Li, Director, Shanghai East Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDGIIIR011
Record Dates: First submitted 2023-08-11; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer; HER2-low-expressing Gastric Cancer
Keywords: HER2-low-expressing
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Disitamab Vedotin and Toripalimab (Experimental): Participants will receive Disitamab Vedotin + Toripalimab every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Disitamab Vedotin; Drug: Toripalimab

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.0mg/kg, intravenously D1, once every 14 days (Q2W)
  Other Names: RC48
Drug: Toripalimab — 3.0 mg/kg, once every 14 days (Q2W)

SUMMARY:
This is a single-arm, prospective, non-randomized, multi-center/single-center, open-label, phase I clinical study aimed at evaluating the efficacy and safety of Disitamab Vedotin in combination with PD-1 as posterior line treatment for patients with advanced HER2-low expressing gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Must voluntarily join this study and sign an informed consent form;
2. Age 18-70 years old (including 18 years old and 70 years old);
3. Expected survival period ≥ 12 weeks;
4. ECOG physical fitness score 0 or 1 point;
5. Patients with incurable and unresectable locally advanced or metastatic gastric cancer (including gastroesophageal junction adenocarcinoma) confirmed by histology or cytology;
6. The HER2 immunohistochemistry (IHC) test results are IHC 1+, the subject's previous test results (confirmed by the investigator) or the test results of the research center are acceptable;
7. The patient has received second-line treatment (at least) after tumor recurrence/metastasis
8. Evidence of tumor disease progression during or after the most recent treatment, as documented by medical history or confirmed by the investigator;
9. At least one measurable lesion according to RECIST 1.1;
10. For female subjects: should be surgically sterilized, postmenopausal patients, or agree to use at least one medically approved contraceptive measure (such as an intrauterine device, contraceptives) during the study treatment period and within 6 months after the end of the study treatment period. pills or condoms), must have a negative blood pregnancy test within 7 days prior to study enrollment, and must be non-lactating; for male subjects: should for surgical sterilization, or agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period of the experimental group subjects;
11. Sufficient organ function:

    1. Bone marrow function: hemoglobin ≥ 9g/dL; absolute neutrophil count ≥ 1.5×109/L; platelet ≥ 100×109/L;
    2. Liver function: serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN); when there is no liver metastasis, alanine aminotransferase (ALT), aspartate aminotransferase (AST and alkaline phosphatase (ALP) ≤ 2.5×ULN, and in the presence of liver metastases ALT, AST, and ALP are ≤ 5×ULN;
    3. Renal function (subject to the normal value of the clinical trial center): blood creatinine ≤ 1.5×ULN, or creatinine clearance rate (CrCl) ≥ 60 mL/min calculated by Cockcroft-Gault formula method, or 24-hour urine CrCl ≥ 60 mL/min;
    4. Heart function: New York Heart Association (NYHA) classification < Grade 3; left ventricular ejection fraction ≥ 50%;
12. Able to understand trial requirements, willing and able to comply with trial and follow-up procedures.

Exclusion Criteria:

1. Brain metastasis or leptomeningeal metastasis;
2. Tumor lesions with a bleeding tendency (e.g., active ulcerated tumor lesions with a positive fecal occult blood test, history of vomiting blood or black stools within 2 months prior to signing the informed consent, risk of gastrointestinal hemorrhage in the judgment of the investigator) or previous blood transfusions in the 4 weeks prior to study drug administration;
3. Suffering from other malignant tumors within 5 years before signing the informed consent form (non-melanoma skin cancer, cervical carcinoma in situ, ductal carcinoma in situ or other tumors that have been effectively treated, except for malignant tumors that are considered cured);
4. Received chemotherapy, radiotherapy, and immune therapy within 4 weeks before the start of the study drug
5. Received palliative radiotherapy for bone metastases within 2 weeks before the start of the study drug;
6. Received anti-tumor traditional Chinese medicine treatment within 2 weeks before the start of the study drug;
7. The toxicity caused by previous anti-tumor therapy has not recovered to CTCAE (version 4.03) grade 0-1 (except for alopecia, hyperpigmentation, and long-term toxicity caused by radiotherapy, which in the judgment of the investigator cannot be recovered);
8. Prior treatment with T-DM1 or participation in a clinical study of this type of drug;
9. The study drug has been used within 4 weeks before the start of the study drug;
10. Major surgery has been performed within 4 weeks before the start of the study drug and the patient has not fully recovered;
11. Have been vaccinated with live vaccines within 4 weeks before the start of the study drug or plan to receive any vaccines during the study period;
12. Arterial/venous thrombotic events, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis, pulmonary embolism, and myocardial infarction, occurred within 1 year before the study drug;
13. Suffering from uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, liver cirrhosis, angina pectoris, serious arrhythmia, etc.;
14. Suffering from active infection requiring systemic treatment;
15. History of active tuberculosis;
16. Positive human immunodeficiency virus (HIV) test result;
17. Patients with active hepatitis B or C (HBsAg positive and HBV DNA titers higher than the upper limit of normal when HBsAg is positive; HCVAb positive and HCV RNA titers higher than the upper limit of normal when HBsAg is positive);
18. Presence of third interstitial fluid that cannot be controlled by drainage or other methods (including massive pleural effusion or ascites);
19. Known to have hypersensitivity or delayed allergic reactions to certain components of RC48-ADC or similar drugs;
20. Exclude, at the investigator's discretion, other conditions that might confuse the study results or affect the subjects' ability to follow the study procedures, such as alcoholism, drug abuse, mental disorders, criminal detention, etc.;
21. Suffering from any other disease, metabolic abnormality, abnormal physical examination, or abnormal laboratory test, according to the judgment of the investigator, there is reason to suspect that the subject has a certain disease or condition that is not suitable for the use of the study drug, or will affect the research results interpretations, or situations that place the subject at high risk;
22. Women who are pregnant or breastfeeding or women/men who are planning to give birth;
23. It is estimated that the subjects' compliance to participate in this clinical study is insufficient or the investigators believe that there are other factors that are not suitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR) per RECIST version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
Overall survival (OS) | 12 months after the last subject participating in
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.
Disease control rate (DCR) | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD)in total subjects
Drug-related safety indicators | 12 months after the last subject participating in
  Exposure to the investigational drug and incidence, nature, and severity of adverse events, including serious adverse events（n, %）

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD,PhD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided